CLINICAL TRIAL: NCT03099252
Title: Caring for Babies: A Study of Ontario Maternal-Newborn Hospitals on the Implementation of Parent-targeted Education (ONesiE)
Brief Title: Caring for Babies: A Study of Ontario Maternal-Newborn Hospitals on the Implementation of Parent-targeted Education
Acronym: ONesiE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Ontario Child Health Support Unit (OCHSU) (Unknown); Better Outcomes Registry & Network Ontario (Unknown); Dalhousie University (Other); Ottawa Hospital Research Institute (Other); University of Calgary (Other); McGill University (Other); The Hospital for Sick Children (Other); Headwaters Health Care Centre (Unknown); Champlain Maternal Newborn Regional Program (Unknown); St Thomas Elgin General Hospital (Unknown); Baby Friendly Hospital Initiative (Unknown)
Responsible Party: Principal Investigator, Denise Harrison, Chair in Nursing Care of Children, Youth and Families, Children's Hospital of Eastern Ontario
Other Study IDs: CHEO REB# 17/01CTO
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled: Participating hospitals will offer the video to all parents on their MBU during the 6 month intervention period (using the preferred delivery methods of the hospital and the parents). The video will be available via multiple means to facilitate optimal parental exposure in diverse settings. This will ensure flexibility of the delivery of the intervention, based on preferences of the nominated nurse leaders and their HCP team, families and available resources.
  All participating maternal/newborn centres will receive the following tools via the designated nurse unit leader of enrolled sites:
  1. Parent-targeted BSweet2Babies video
  2. Parent cards- Reminder for parents of video, with Quick Response (QR) code of the video
  3. BSweet2Babies Poster-visual reminder for parents and HCP's on the enrolled units
  4. Monthly support calls for the nursing leaders of the Mother Baby Units (MBU)
  5. Bi-monthly community of practice teleconferences for the nursing leaders of the MBU
  Interventions: Other: Parent-targeted BSweet2Babies video

INTERVENTIONS:
Other: Parent-targeted BSweet2Babies video — The video portrays three babies having blood tests while being i) BF, ii) held SSC with the mother, and iii) receiving sucrose. The calming effects of these strategies are powerfully portrayed. Voice-over in user-friendly language explains how parents can help their babies by partnering with clinicians to use these strategies. As per the definition of patient-targeted and mediated interventions, this video is: i) patient (parent)-targeted, as it actively engages parents to improve their knowledge, positively affect their experience (during newborn screening), change their behavior and their baby's outcomes; ii) patient-mediated, as the video enables parents to change health professional behavior.

SUMMARY:
Newborn infants have blood work procedures for newborn screening and bilirubin testing in their first days of life that cause pain, distress and physiological changes. Breastfeeding (BF), skin to skin care (SSC), or giving small amounts of sweet solutions (sucrose or glucose) with or without a pacifier, effectively and safely reduce pain and distress in newborn infants during painful procedures. However, studies of neonatal pain management practices in Ontario and throughout Canada demonstrate inconsistent use of these strategies. There is a clear need for developing and testing acceptable parent-targeted interventions, alongside health care provider (HCP)-targeted knowledge translation (KT) interventions, to support parents' involvement in comforting their infants during painful procedures. To address this knowledge to action (KTA) gap, Denise Harrison's Be Sweet to Babies team developed the BSweet2Babies video, which demonstrates the effectiveness of BF, SSC, and sucrose during infant bloodwork and how parents can use and advocate for these pain management strategies.

This project addresses a knowledge to practice gap that is highly relevant to all babies and their families. Thus, this study has the potential to advance health care of all babies and contribute to the science of KT by evaluating the implementation of a parent-targeted and mediated KT strategy in diverse hospital settings.

Hospitals were eligible for inclusion if they (1) provide Level 1 or Level 2 maternal/newborn care contributing data to the Better Outcomes Registry & Network Ontario (BORN) Information Systems (BIS); (2) have a birth volume of at least 50 per year; (3) have <85% use of pain management (BF,SSC, sucrose) during newborn screening or bilirubin sampling, as per BIS data; and (4) have < 50% missing data for the pain management data element in the BIS. Participating hospitals will receive a tablet and will offer all parents the 5 minute BSweet2Babies video before newborn bloodwork. BORN Information System (BIS) data will subsequently be analyzed to evaluate the use of BF, SSC and sweet solutions.

DETAILED DESCRIPTION:
Background: Newborn infants have blood work procedures for newborn screening and bilirubin testing in their first days of life that cause pain, distress and physiological changes. Breastfeeding (BF), skin to skin care (SSC), or giving small amounts of sweet solutions (sucrose or glucose) with or without a pacifier, effectively and safely reduce pain and distress in newborn infants during painful procedures. However, studies of neonatal pain management practices in Ontario and throughout Canada demonstrate inconsistent use of these strategies. There is a clear need for developing and testing acceptable parent-targeted interventions, alongside health care provider-targeted knowledge translation (KT) interventions, to support parents' involvement in comforting their infants during painful procedures. To address this knowledge to action (KTA) gap, Denise Harrison's Be Sweet to Babies team developed the BSweet2Babies video, which demonstrates the effectiveness of BF, SSC, and sucrose during infant bloodwork and how parents can use and advocate for these pain management strategies.

Objectives: To conduct a process evaluation to understand during the 6-month intervention period; (1) to what extent did HCPs implement the BSweet2Babies video in their setting; (2) What were the barriers and facilitators encountered in implementing the BSweet2Babies video; (3) What were the barriers and facilitators encountered in implementing the evidence shown in the BSweet2babies video (i.e. breastfeeding, skin-to-skin care, sucrose).

Study design and methods: Sequential exploratory mixed methods study. The mixed methods implementation study includes process evaluation, exploration of facilitators and barriers to implementation of the video and uptake of the demonstrated recommended pain management of BF, SSC or sucrose during initial blood sampling by heel prick.

Data Analysis: Directed content analysis will be used to analyse the qualitative data (i.e. monthly phone calls and bi-monthly community of practice teleconferences). Interview data will be transcribed verbatim with consent. A deductive and inductive approach will be used to code the qualitative data with codes developed apriori based on the Theoretical Domains Framework. Any concepts that do not fit within the framework will be assigned a new code.

Process evaluation will be described and summarized according to the process evaluation of complex intervention guide.

BORN Ontario data analysts in consultation with CoI Taljaard will conduct analysis using descriptive statistics to compare characteristics of participating sites and births including unit type (Level 1 compared to Level 2), birth volume, infant sex, and parity. In addition, BIS pain data will be reported as baseline and following the 6- month implementation period.

ELIGIBILITY:
Inclusion criteria for hospitals include:

* Hospitals providing Level 1 and Level 2 maternal/newborn care contributing data to the BIS
* A birth volume of at least 50 per year

Hospitals will be excluded if they:

* >85% use of pain management (BF, SSC, sucrose) during newborn screening
* >50% missing data for the pain management data element in the BIS. element.
* two hospitals that were used as pilot sites will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Ontario hospitals that provide Level 1 or Level 2 maternal/newborn care, contributing data to the BORN Information System and meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Process Evaluation | 7 months.
  Directed content analysis will be used to analyze data from monthly interview, bi-monthly teleconferences and end of intervention surveys
BORN BIS Pain Data | Six months prior to study launch date.
  Number of effective pain treatment used during newborn screening.
BORN BIS Pain Data | Six months following completion of the intervention.
  Number of effective pain treatment used during newborn screening.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Harrison, RN, PhD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No